CLINICAL TRIAL: NCT05348720
Title: Impact of a COVID-19 Related ICU Stay on Mental Health for Patients and Their Relatives. An Exploratory 18-month Follow-up Study for COVID-19 ICU Survivors and Their Relatives.
Brief Title: Impact of a COVID-19 Related ICU Stay on Mental Health for Patients and Their Relatives
Acronym: PICOVIDS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Stoffel Lamote, Medical Doctor, Intensive Care Unit, General Hospital Groeninge
Other Study IDs: AZGS2021059
Record Dates: First submitted 2022-04-15; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Post Intensive Care Syndrome; PICS; COVID-19; Critically Ill; Mental Health
Keywords: COVID-19; ICU survivor; PICS; PICS-F; neurocognitive sequels; Follow-up
MeSH Terms: conditions — postintensive care syndrome; COVID-19; Critical Illness; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 ICU survivor: COVID-19 patients admitted to ICU between the 1st of March 2020 and the 30rd of May 2021, who survived ICU stay and still alive 18 months after ICU discharge.
- Relatives: Relative of those COVID-19 patients enrolled in the 'COVID-19 ICU survivor' cohort

SUMMARY:
As ICU mortality has been significantly decreased over the last two decades, the focus has been shifting from short term (such as ICU and hospital mortality) to long-term outcome. This evolution has led to a new entity that has been established in 2012 at a stakeholder conference: the Post-Intensive Care Syndrome (PICS). It is defined as impairments in physical, cognitive and mental health status arising after critical illness and persisting beyond acute care hospitalisation. As family members of ICU patients may also be affected by mental health impairment, the PICS-F (F for Family) has been introduced simultaneously.

It is expected that the COVID-19 pandemic will result in a significant increase of the proportion of patients and relatives suffering PICS and PICS-F, as there is during the COVID-19 related ICU-stay exposure to a high number of risk factors for developing these entities.

This Post Intensive Care Syndrome in COVID-19 survivors (PICOVIDS) study is an observational, single-center exploratory follow-up cohort study that aims to get insight into the mental impact of a COVID-19 related ICU stay for COVID-19 ICU survivors and their family members, 18 months after ICU discharge.

Specific research questions are:

1. What is the prevalence of symptoms of depression, anxiety and Post Traumatic Stress Disorder (PTSD) and what is the prevalence of these specific disorders in COVID-19 ICU-survivors and their relatives 18 months after ICU-discharge?
2. What are important risk factors for these symptoms and disorders?
3. What is the satisfaction level of patient and caregiver about the ICU care: How did they experience ICU stay?

DETAILED DESCRIPTION:
Design:

The Post Intensive Care Syndrome in COVID-19 survivors (PICOVIDS) study is an observational, single-center exploratory follow-up cohort study in a non-university hospital with 31 ICU beds.

Objective:

The study aims to get insight into the mental impact of a COVID-19 related ICU stay for COVID-19 ICU survivors and their family members, 18 months after ICU discharge.

Specific research questions are:

1. What is the prevalence of symptoms of depression, anxiety and Post Traumatic Stress Disorder (PTSD) and what is the prevalence of these specific disorders in COVID-19 ICU-survivors and their relatives 18 months after ICU-discharge?
2. What are important risk factors for these symptoms and these disorders?
3. What is the satisfaction level of patient and caregiver about the ICU care: How did they experience ICU stay?

Patients' recruitment (See section 'inclusion and exclusion criteria' for further details):

Patients admitted to the ICU between 1 March 2020 and 31 May 2021, with respiratory failure primarily due to COVID-19, who survived ICU stay and hospitalisation are eligible and will be contacted by telephone 16 to 18 months after ICU discharge by the research team. Patients will receive information regarding the aim, content and relevance of the study and asked for participation to this study. They will be asked as well whether his or her caregiver the most involved during the ICU stay would participate to the study.

Methods:

Once oral informed consent by telephone will be given, a bundle will be sent to patient and involved relative by post. This bundle contains informed consent, information brochure and several questionnaires.

Questionnaires for patients are:

* Hospital and Depression Scale (HADS anxiety and depression)
* Patient Checklist for DSM-5 (PCL-5) for COVID
* Cognitive Failure Questionnaire (CFQ)
* Short Form 36 Health Survey Questionnaire (SF-36)
* Questionnaire for persistent physical complaints
* Rockwood Clinical Frailty Scale
* Patient Continuity of Care Questionnaire adjusted (PCCQ): subscales relationship in hospital, information transfer)
* Socio-demographic questionnaire

Caregivers will receive the same questionnaires except for the SF-36, the questionnaire assessing persistent physical complaints and the Rockwood Clinical Frailty Scale as these one are not applicable to them, while a Caregiver Reaction Assessment (CRA) scale questionnaire will be added for this cohort.

Consequently psychological, cognitive and physical symptoms, clinical frailty, satisfaction level about care and socio-demographic factors will be assessed.

There are Dutch, French and English versions of this bundle available, as preferred by patient and relative.

Patient and caregiver will be contacted a second time by telephone 10 to 14 days after the first call for verifying whether there are remaining questions after receiving the bundle. A second bundle will be sent by post in case of the first one would have been lost or patient and/or caregiver couldn't be reached.

Questionnaires will be analysed by two members of the research team. Patients and caregivers scoring more than 7 on the HADS-Anxiety, more than 8 on the HADS-Depression or more than 32 on the PCL-5 COVID questionnaire will be considered as having symptoms of respectively anxiety, depression and PTSD. Subsequently, they will be invited for a clinical and structured interview, using the Mini-International Neuropsychiatric Interview (MINI), the Clinician-Administered PTSD scale (CAPS) and the Montreal cognitive Assessment (MoCa). A psychiatrist and clinical psychologist will conduct this interview. Consequently, diagnosis of Generalised Anxiety Disorder (GAD), Depression and PTSD according to the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) as well as cognitive impairment could be established.

Data Collection:

On the one hand, anonymised patient data with respect to the ICU hospitalisation will be collected from patient records (electronic patient records, Patient Data Management System (PDMS), Klinisch Werkstation (KWS), Cyberlab). This data collecting process will be facilitated by LynxCare® company, an Artificial Intelligence (AI) and Natural Language Processing (NLP) based big data platform. This medical data will include: demographics, pre-existing co-morbidities (including Clinical Frailty score (CFS) and Charlson Comorbidity Index, severity of illness scores (APACHE-II score, Simplified Acute Physiology Score (SAPS), Sequential Organ Failure Assessment (SOFA)), specific COVID-treatment, method of respiratory support during ICU stay (High Flow Oxygen, Non-Invasive Ventilation, Mechanical Ventilation, prone ventilation, Extracorporeal Membrane Oxygenation (ECMO), duration of mechanical ventilation, duration of ECMO run, diagnosis of ICU-Acquired Weakness (ICU-AW) or Critical Illness Polyneuropathy (CIP) and Myopathy (CIM, presentation of Acute Kidney Injury (AKI) grade 3 of need for dialysis, ICU-Length of stay (LOS), Hospital-LOS Additionally, specific interest will go to data regarding potential risk factors for long-term neurocognitive sequels such as: age, social context, pre-existing psychiatric and/or cognitive symptoms, neurological events during ICU hospitalisation (e.g. delirium, ICU-AW, CIP and CIM, stroke (ischemic or hemorrhagic)), need for mechanical ventilation, need for ECMO, need for multiple sedative agents, AKI with or without need for dialysis, ICU-LOS, hospital-LOS, persisting symptoms after discharge, duration of work-related problems (duration of sick leave), increased dependence after discharge, inability to return to original home situation, loss of other family members during follow-up period.

On the other hand, data about long-term outcome will be collected from questionnaires and a possibly clinical interview (for details with regards to this data: see section 'methods').

Data analysis Data will be merged ad patient level. Descriptive statistics will be used to describe baseline characteristics, inpatient course during index hospitalisation and findings (prevalence of the various long-term outcome) obtained from the questionnaires for patient and relatives. Regression analysis will be used to determine associations between patient characteristics, inpatient course and long-term outcomes.

Software Package for the Social Sciences (SPSS) will be used for data analysis.

Data management and ethical considerations Both data extracted from medical records and from the questionnaires will be anonymised before analysis and will be merged at patient level. Data management will be performed by the team of Lynxcare® and by the research team (study nurses and investigators).

Importantly, LynxCare® will only have access to the encrypted data, only the research team will have the key for decoding. This all will be strictly conform the most recent European Union's General Data Protection Regulation (GDPR). Hence patient's privacy will be guaranteed maximally throughout the whole process.

Patients will be asked for oral informed consent during the first phone call, followed by obtaining a written informed consent for both patient and relative, a form that will be included in the bundle sent by post. This written (signed) informed consent is a strict condition prior to enrollment, data collection and analysis.

Ethical approval was given by the Medical Ethical Committee AZ Groeninge (B3962021000047), all patients will give their informed consent prior to data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patient admitted to the ICU between 1st of March 2020 and 31st of May 2021
* Surviving ICU and index hospitalisation
* Respiratory failure due to COVID-19 with need for High Flow Oxygen Therapy (HFOT), non-invasive ventilation (NIV) or mechanical ventilation (MV)
* Family member (caregiver) of eligible COVID-19
* Written informed consent obtained from patient and family member

Exclusion Criteria:

* ICU length of stay (ICU-LOS) </= 72h
* Decease of the COVID-19 patient during 18-month follow-up period
* Respiratory failure and admission to ICU was not primary related to COVID-19
* Poor or moderate knowledge of Dutch, French or English language
* Mentally not able to complete questionnaires or to give informed consent, due to a neurocognitive deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COVID-19 patients admitted to the ICU between 1/3/2020 and 31/5/2021, who survived the ICU and index hospitalisation, requiring High Flow Oxygen Therapy (HFOT), non-invasive ventilation (NIV) or mechanical ventilation (MV) due to respiratory failure primarily related to COVID-19, will be eligible.
  Covid-19 diagnosis will be based on RNA detection of SARS-COV-2 using RT-PCR of a nasopharyngeal swab or through respiratory specimen obtained by bronchoscopy.
  All eligible patients, still alive 18 months after ICU discharge, will be contacted by telephone for participation in this study. Simultaneously, these patients will be asked if their family member is keen to participate in the study as well. We aim to enroll the family member the most involved in the patient's ICU stay.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: Prevalence of psychiatric symptoms in COVID-19 ICU survivors | 18 months after ICU discharge
  symptoms of anxiety(1), depression(2) and PTSD(3) (1+2) anxiety and depression measured using the HADS symptom score (score range 0 (best) to 42 (worst)): presence of symptoms of anxiety if HADS anxiety subscale > 7; presence of symptoms of depression if HADS depression subscale > 8; (3) presence of PTSD-related symptoms measured using the PCL-5 COVID score (score range 17 (not all PTSD) to 85(most extreme form of PTSD): PTSD symptoms if score > 32.
Composite outcome: Prevalence of psychiatric symptoms among relatives of COVID-19 ICU survivors | 18 months after ICU discharge
  symptoms of anxiety(1), depression(2) and PTSD(3) (1+2) anxiety and depression measured using the HADS symptom score (score range 0 (best) to 42 (worst)): presence of symptoms of anxiety if HADS anxiety subscale > 7; presence of symptoms of depression if HADS depression subscale > 8; (3) presence of PTSD-related symptoms measured using the PCL-5 COVID score (score range 17 (not all PTSD) to 85(most extreme form of PTSD): PTSD symptoms if score > 32.

SECONDARY OUTCOMES:
Composite outcome: Prevalence of psychiatric disorders among relatives of COVID ICU survivors. | 18 months after ICU discharge
  Assessed during clinical interview. Generalised Anxiety Disorder (GAD) and depression using DSM-5 criteria as assessed in Mini-International Neuropsychiatric Interview (MINI). PTSD as assessed using Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
Composite outcome: Prevalence of psychiatric disorders among COVID ICU survivors. | 18 months after ICU discharge
  Assessed during clinical interview. Generalised Anxiety Disorder (GAD) and depression using DSM-5 criteria as assessed in Mini-International Neuropsychiatric Interview (MINI). PTSD as assessed using Clinician Administered PTSD Scale for DSM-5 (CAPS-5).
Prevalence of cognitive impairment in COVID-19 ICU survivors and their relatives | 18 months after ICU discharge
  Cognitive Failure Questionnaire (CFQ) with score ranging from 0 (no impairment) to 100 (maximum impairment)
Impact of caring for COVID-19 ICU survivor after hospital discharge on the relative | 18 months after ICU discharge
  Caregiver Reaction Assessment (CRA) scale for relatives: multidimensional measure of the reaction of the relative to caring for a COVID-19 ICU survivor after hospital discharge. Evaluation by 5 point Likert scale (ranging from 1 = strongly disagree to 5 = strongly agree). Domains assessed are financial problems, disrupted schedule, lack of family support, health problems and self-esteem.
Patient and relatives' satisfaction level about continuity of care after hospital discharge | 18 months after ICU discharge
  Patient Continuity of Care Questionnaire adjusted (PCCQ) for both patient and relative: total score of the questionnaire ranges from 6 to 30, higher score indicates higher continuity while a score < 24 indicates insufficient continuity.

CONTACTS AND LOCATIONS:
Overall Officials: Stoffel Lamote, MD, Principal Investigator — General Hospital Groeninge
Locations (1):
- AZ Groeninge Kortrijk, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Gulati A, Pomeranz C, Qamar Z, Thomas S, Frisch D, George G, Summer R, DeSimone J, Sundaram B. A Comprehensive Review of Manifestations of Novel Coronaviruses in the Context of Deadly COVID-19 Global Pandemic. Am J Med Sci. 2020 Jul;360(1):5-34. doi: 10.1016/j.amjms.2020.05.006. Epub 2020 May 11. PMID 32620220
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Writing Committee for the COMEBAC Study Group; Morin L, Savale L, Pham T, Colle R, Figueiredo S, Harrois A, Gasnier M, Lecoq AL, Meyrignac O, Noel N, Baudry E, Bellin MF, Beurnier A, Choucha W, Corruble E, Dortet L, Hardy-Leger I, Radiguer F, Sportouch S, Verny C, Wyplosz B, Zaidan M, Becquemont L, Montani D, Monnet X. Four-Month Clinical Status of a Cohort of Patients After Hospitalization for COVID-19. JAMA. 2021 Apr 20;325(15):1525-1534. doi: 10.1001/jama.2021.3331. PMID 33729425
- [Background] Taquet M, Geddes JR, Husain M, Luciano S, Harrison PJ. 6-month neurological and psychiatric outcomes in 236 379 survivors of COVID-19: a retrospective cohort study using electronic health records. Lancet Psychiatry. 2021 May;8(5):416-427. doi: 10.1016/S2215-0366(21)00084-5. Epub 2021 Apr 6. PMID 33836148
- [Background] Jaffri A, Jaffri UA. Post-Intensive care syndrome and COVID-19: crisis after a crisis? Heart Lung. 2020 Nov-Dec;49(6):883-884. doi: 10.1016/j.hrtlng.2020.06.006. Epub 2020 Jun 18. No abstract available. PMID 32690219
- [Background] Herridge MS, Moss M, Hough CL, Hopkins RO, Rice TW, Bienvenu OJ, Azoulay E. Recovery and outcomes after the acute respiratory distress syndrome (ARDS) in patients and their family caregivers. Intensive Care Med. 2016 May;42(5):725-738. doi: 10.1007/s00134-016-4321-8. Epub 2016 Mar 30. PMID 27025938
- [Background] Cameron JI, Chu LM, Matte A, Tomlinson G, Chan L, Thomas C, Friedrich JO, Mehta S, Lamontagne F, Levasseur M, Ferguson ND, Adhikari NK, Rudkowski JC, Meggison H, Skrobik Y, Flannery J, Bayley M, Batt J, dos Santos C, Abbey SE, Tan A, Lo V, Mathur S, Parotto M, Morris D, Flockhart L, Fan E, Lee CM, Wilcox ME, Ayas N, Choong K, Fowler R, Scales DC, Sinuff T, Cuthbertson BH, Rose L, Robles P, Burns S, Cypel M, Singer L, Chaparro C, Chow CW, Keshavjee S, Brochard L, Hebert P, Slutsky AS, Marshall JC, Cook D, Herridge MS; RECOVER Program Investigators (Phase 1: towards RECOVER); Canadian Critical Care Trials Group. One-Year Outcomes in Caregivers of Critically Ill Patients. N Engl J Med. 2016 May 12;374(19):1831-41. doi: 10.1056/NEJMoa1511160. PMID 27168433
- [Background] van Beusekom I, Bakhshi-Raiez F, de Keizer NF, Dongelmans DA, van der Schaaf M. Reported burden on informal caregivers of ICU survivors: a literature review. Crit Care. 2016 Jan 21;20:16. doi: 10.1186/s13054-016-1185-9. PMID 26792081
- [Background] Azoulay E, Resche-Rigon M, Megarbane B, Reuter D, Labbe V, Cariou A, Geri G, Van der Meersch G, Kouatchet A, Guisset O, Bruneel F, Reignier J, Souppart V, Barbier F, Argaud L, Quenot JP, Papazian L, Guidet B, Thiery G, Klouche K, Lesieur O, Demoule A, Guitton C, Capellier G, Mourvillier B, Biard L, Pochard F, Kentish-Barnes N. Association of COVID-19 Acute Respiratory Distress Syndrome With Symptoms of Posttraumatic Stress Disorder in Family Members After ICU Discharge. JAMA. 2022 Mar 15;327(11):1042-1050. doi: 10.1001/jama.2022.2017. PMID 35179564
- [Background] Heesakkers H, van der Hoeven JG, Corsten S, Janssen I, Ewalds E, Simons KS, Westerhof B, Rettig TCD, Jacobs C, van Santen S, Slooter AJC, van der Woude MCE, van den Boogaard M, Zegers M. Clinical Outcomes Among Patients With 1-Year Survival Following Intensive Care Unit Treatment for COVID-19. JAMA. 2022 Feb 8;327(6):559-565. doi: 10.1001/jama.2022.0040. PMID 35072716
- [Background] van Veenendaal N, van der Meulen IC, Onrust M, Paans W, Dieperink W, van der Voort PHJ. Six-Month Outcomes in COVID-19 ICU Patients and Their Family Members: A Prospective Cohort Study. Healthcare (Basel). 2021 Jul 8;9(7):865. doi: 10.3390/healthcare9070865. PMID 34356243